CLINICAL TRIAL: NCT02400489
Title: Clinical Study to Evaluate the Performance of Perimount Heart Valve in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Perimount CN001
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Mitral Valve or Aortic Valve Replacement
Keywords: Heart Valve Replacement Surgery; Perimount; Edwards

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
To recruit patients who implanted with Perimount Heart Valve (Type Number: 6900PTFX or 2800TFX) from three hospitals in China.

To track the patients'situations during one year after surgery and to collect the relevant clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with Perimount 6900PTFX after 2012-11-19 or with Perimount 2800TFX after 2013-8-20
* Patients sign the Inform Consent Form (ICF) and agree to join the study

Exclusion Criteria:

* Don't have any specific exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with Perimount 6900PTFX or Perimount 2800TFX in three hospitals in China: Wuhan Asia Heart Hospital, Shandong Provincial Hospital, Tianjin Chest Hospital.
  Patients need to complete two follow up visits after surgery in hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Twice echocardiography to evaluate the performance of heart valve | Compare the 1st echocardiography at average 6 months after surgery and 2nd echocardiography at 12 months after surgery
  subjects need to do the echocardiography in two follow up visits
The recovery status of patients after surgery | The subjects will be followed for the duration of one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xufa Chen, M.D, Principal Investigator — Wuhan Asia Heart Hospital; Chengwei Zou, M.D, Principal Investigator — Shandong Provincial Hospital; Nan Jiang, M.D, Principal Investigator — Tianjin Chest Hospital
Locations (3):
- China (3):
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Shandong Provincial Hospital, Jinan, Shandong
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.